CLINICAL TRIAL: NCT01364753
Title: Age-related Longitudinal Changes in Aviator Performance
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jerome A Yesavage,, Professor, Stanford University
Other Study IDs: SU-06302009-2940; R37AG012713 (NIH)
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Memory Impairment
Keywords: Memory; Aviation
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pilots: No intervention; observational study

SUMMARY:
Our overall goal has been twofold: 1) to evaluate whether there are significant age-related changes in flight simulator performance near age 60, and 2) to assess whether there is an alternative model that can explain longitudinal flight simulator performance on the basis of measures of cognitive function and expertise.

DETAILED DESCRIPTION:
Our overall goal has been twofold: 1) to evaluate whether there are significant age-related changes in flight simulator performance near age 60, and 2) to assess whether there is an alternative model that can explain longitudinal flight simulator performance on the basis of measures of cognitive function and expertise. Such a model might be able to predict change in aviator performance better than what could be predicted by chronological age alone.

ELIGIBILITY:
Inclusion Criteria:1) licensed aircraft pilot 2) 45 to 70 years of age 3) at least 100 hours of total flight experience 4) current FAA (Federal Aviation Administration) medical certificate of class III or higher

Exclusion Criteria:1) taking psychotropic medications 2) taking other medications with arousal or sedative effects

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy older pilots holding active airplane license
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2006-01; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Aviation-related performance over time. | longitudinal
  Participants "fly" in our computerized flight simulator and perform a set of brief tasks designed to measure reaction time and attention span. The study is longitudinal, collecting information about aviation-related performance over time. There is an initial training period, followed by annual visits. During the training period participants learn how to "fly" the simulator, and performance on certain standard maneuvers will be measured during a maximum of 6 simulated flights. At each annual visit, participants fly two 75-minute simulated flights and may be asked to perform up to four holding patterns and instrument landings.

CONTACTS AND LOCATIONS:
Overall Officials: Jerome A Yesavage, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States